CLINICAL TRIAL: NCT06039852
Title: Breathe-Easy: a Pilot Study to Examine the Acceptability and Feasibility of a Novel Postural Management Night-time Intervention to Improve Respiratory Health of Children With Complex Neuro-disability.
Brief Title: Acceptability and Feasibility of a New Postural Management Night-time Intervention to Improve Respiratory Health of Children With Complex Neuro-disability
Acronym: Breathe-Easy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sussex Community NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 288217
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Aspiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Novel Postural Management Night-time Intervention Components (Experimental): Intervention Arm
  Interventions: Other: Novel Postural Management Night-time Intervention

INTERVENTIONS:
Other: Novel Postural Management Night-time Intervention — Essential elements and components of PMN-TI:
  * Safe and comfortable position to enable sleep
  * Positioning to enable UAD overnight
  * Quiet breathing unobstructed by base of tongue (i.e. stertor), vocal cords (i.e. stridor) or pooled secretions
  * Postural support in lying to achieve comfort, promote symmetry of posture and maximum loadbearing
  * Stomach contents reduced or emptied overnight to minimize reflux and associated aspiration risk.

SUMMARY:
This research concerns children with complex neuro-disability. Damage to the developing brain leads to lifelong disturbances in motor control, seizures, cognition, communication, eating and drinking, and behaviour. Children with complex neuro-disability are dependent upon others to move and position them. Children commonly experience chronic lung disease, leading to frequent hospitalisation, medical interventions and premature death. Respiratory illness may be triggered by "aspiration", i.e. when saliva, food, liquid or stomach contents enter the lungs. Aspiration risks increase at night-time when supervision is limited and children are positioned on their backs. Some children experience repeated breathing complications requiring prolonged hospital stays including respiratory support in intensive care.

Consultant Respiratory Paediatrician Akshat Kapur and Physiotherapist Hilda Perry developed a new night-time intervention to improve respiratory health of children with complex neuro-disability. Dr Kapur and his team have found that this intervention can help reduce respiratory illness and time spent in hospital for some children. This is an acceptability and feasibility study which means the investigators want to find out if this new intervention is something that children with complex neuro-disability and their families are happy (i.e. it is acceptable) and able (i.e. it is feasible) to do. If so, a larger future research study can be designed to find out if the intervention works to improve the respiratory health of children with complex neuro-disability.

DETAILED DESCRIPTION:
The intervention involves positioning children safely on their fronts using pillows to support the body under the shoulder and hip, and with the head slightly lowered so that gravity can help drain secretions from the mouth. This is different to current night-time positioning recommendations of either lying children on their backs or side. The new intervention also involves, where possible, the draining of children's stomach contents overnight via an existing feeding tube to prevent aspiration of stomach contents.

The investigators will work closely with 10 children with complex neuro-disability and their families, and health professionals as investigators introduce this new night-time intervention. The investigators will make observations about children's respiratory and sleep outcomes before and after making changes. The investigators will make comparisons using questionnaires, sleep diaries, records of antibiotic use and hospital admissions. The investigators will collect this information before making any changes, at 3 months after the intervention has been established and after 6 months when the study ends. The investigators will talk to children, parents, carers and relevant health professionals to find out what they think and feel about the new intervention, including any issues/challenges that occurred.

The investigators will record how many children and families were approached to take part in the study. The investigators will record how many agreed to take part, how many chose to leave half way through and how many said they did not want to take part in the study. Families who discontinued or who declined the intervention will be given opportunity to provide feedback confidentially.

The investigators will use the findings to decide whether it is feasible and acceptable to children and families to run a research trial of this new night-time intervention. The data will help us to design a future research trial.

ELIGIBILITY:
Inclusion Criteria:

* dependent upon others to position/move their bodies
* high risk of aspiration linked to swallowing difficulties
* aged 2-18yrs
* have gastrostomy/jejunostomy
* receiving care from Consultant Respiratory Paediatrician from Royal Alexandra Children's Hospital (Dr Kapur or colleague) because of recent history of chest infections.

Exclusion Criteria:

* Children with complex neuro-disability who cannot be positioned in such a way that promotes upper airway drainage
* Children using a naso-gastric tube
* Children who do not have a gastrostomy or jejunostomy

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Liverpool Respiratory Symptom Questionnaire | 2 years
  Questionnaire Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Crombie, PhD, Principal Investigator — Sussex Community NHS FT
Locations (1):
- Chailey Clinical Services, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No